CLINICAL TRIAL: NCT04111900
Title: Effect of Sleep on the Recovery of Patients Admitted to the ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16111002
Record Dates: First submitted 2019-09-09; First posted 2019-10-01 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Critical Illness; Circadian Dysregulation; Delirium
MeSH Terms: conditions — Critical Illness; Chronobiology Disorders; Delirium | interventions — Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep/Circadian Friendly (Experimental): initiation of sleep/circadian rhythm friendly intervention the first night spent in MICU after enrollment until patient transfers/discharges, ceases participation, or meets exclusion criteria.
  Interventions: Behavioral: Sleep/Circadian Friendly
- Usual Care (No Intervention): Usual care within intensive care unit

INTERVENTIONS:
Behavioral: Sleep/Circadian Friendly — This intervention attempts to improve sleep and prevent circadian rhythm dysregulation among patients admitted to the medical intensive care unit (MICU). Patients within his arm will be asked to try to keep their TV off and limit their telephone use from 10pm-7am, as well as limit the amount of visitors in their room as much as possible between those hours. Patients will also be offered ear plugs and eye masks if they wish to use at night to aid in helping them sleep, if deemed medically safe to do so. Additionally nurses will be asked to bathe patients either before 10pm or after 7am, to limit their conversations in the patient's room at night, and try as much as possible to limit blood draws and waking patients during those hours as is medically safe. Nurses will also be instructed to lower the blinds in the room at 10 pm and raise them up at 7am to help with patients sleep/wake cycle.
  Arms: Sleep/Circadian Friendly

SUMMARY:
The investigators plan to create several sleep/circadian rhythm friendly rooms within the medical intensive care unit to determine if decreasing sleep fragmentation effects recovery in patients hospitalized in the ICU.

DETAILED DESCRIPTION:
Critically ill patients are known to suffer from severely fragmented sleep with a predominance of stage I sleep and a paucity of slow wave and REM sleep. The causes of this sleep disruption include the intensive care unit (ICU) environment, medical illness, psychological stress, and many of the medications and other treatments used to help those who are critically ill. Surveys have identified poor sleep as one of the most frequent complaints among patients who have survived a critical illness. Patients in medical, cardiac, and surgical ICUs almost uniformly have fragmented sleep.

Although illness, pain, and medications contribute to sleep disruption in ICU patients, the primary factor causing sleep disruption had been thought to be the ICU environment. Noise from various sources, including ventilators, alarms, television, phones, beepers, and conversation, have all been purported to disturb sleep in the ICU. Patients have reported that noise, specifically talking, is a frequent cause of sleep disruption in the ICU. Several studies have confirmed that peak noise levels in ICUs are far in excess of 45 dB during the day and 35 dB at night, which are the recommendations of the Environmental Protection Agency for peak noise levels in the ICU.

The clinical importance of this type of sleep disruption in critically ill patients, however, is not known. The investigators hope to determine if placing patients in sleep/circadian rhythm friendly rooms will enable them to achieve better sleep, suffer from decreased delirium, and have improved recovery from their critical illness.

ELIGIBILITY:
Inclusion Criteria:

* any adult patient admitted to the MICU with an expected length of stay of at least 3 days

Exclusion Criteria:

* frequent overnight neurological checks or frequent peripheral vascular checks

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Length of Stay in ICU | through study completion, an average of 3-4 days
  Time spent from admission to ICU until transfer/discharge or study cessation
Overall Hospital Length of Stay | at study completion, an average of 5-7 days
  Total time spent from admission to ICU until discharge from hospital
Rate of ICU mortality | at study completion, up to 30 days
  rate of mortality while admitted to ICU
Rate of Delirium | Once daily throughout study, on average 3-4 days
  Assess development of delirium through administration of CAM-ICU and RASS performed daily by nursing staff per routine care. Delirium will be considered present if CAM-ICU is positive or RASS above +1 or below -1 at anytime during study.
Hospital Readmission Rate | 30 days after discharge
  rate of hospital readmission within 30-days of discharge

SECONDARY OUTCOMES:
ICU sleep score | daily through study completion, an average of 3-4 days
  Assess sleep quality through administration of Richard Campbell Sleep Questionnaire (RCSQ). RCSQ is a simple and validated survey to measure sleep quality in ICU settings. RCSQ consists of a series of 8 patient reported questions covering sleep depth, sleep latency, total amount of sleep, number of awakenings, sleep quality, noise rating, light rating, and sleep quality compared to at home. All questions are to be reported on a scale of 0-100 with higher values corresponding to better sleep values.
Overnight Sound Intensity Levels | through study completion, an average of 3-4 days
  sound intensity (decibel) within patient room with be continuously recorded through SDL-600 industrial decibel monitors.
Overnight Light Intensity Exposure | through study completion, an average of 3-4 days
  amount of light patients are exposed to overnight, measured in lux, will be continuously recorded through specialized medical lux monitors.
Concentration of Interleukin-6 (IL-6) and interleukin-10 (IL-10) | Study Day 1 and Day 2
  concentrations of IL-6 (pg/mL) and IL-10 (pg/mL), inflammatory cytokines found to play a role in circadian regulation, levels will be measured from approximately 2mL of plasma that will be collected concurrently during morning routine care lab draw.
Concentration of 6-sulphatoxymelatonin (aMT6s) | Study Day 1 and Day 2
  concentrations of 6-sulphatoxymelatonin (pg/mL), the primary urine metabolite of melatonin and circadian rhythm phase marker, will be measured from left-over voided urine collected from patients prior to discard.
Concentration of Lipopolysaccharide binding protein (LBP) | Study Day 1 and Day 2
  Levels of LBP (pg/mL), an acute phase protein that upregulates during an inflammatory physiologic state, will be measured from 2mL of blood taken concurrently with routine morning labs.

CONTACTS AND LOCATIONS:
Overall Officials: Garth R Swanson, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States